CLINICAL TRIAL: NCT04814745
Title: Intrathecal Morphine Compared to Intravenous Tramadol and Transversus Abdominal Plane Block for Catheter Related Bladder Discomfort Syndrome
Brief Title: Intrathecal Morphine for Radical Robot Assisted Prostatectomy (TORNADO)
Acronym: TORNADO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3236
Record Dates: First submitted 2021-01-15; First posted 2021-03-24 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Catheter Related Complication
MeSH Terms: interventions — Morphine; Infusions, Intravenous; Tramadol; Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- morphine (Active Comparator): morphine 150 mcg will be administered intrathecally before surgery by using a 25 Gauge with acre spinal needle
  Interventions: Drug: intrathecal infusion
- tramadol (Active Comparator): tramadol 400 mg will be administered by using an elastomeric pump for 24 hours after surgery
  Interventions: Drug: Intravenous Infusion
- ropivacaine (Active Comparator): at the end of surgery transversus abdominis plane block will be performed bilaterally and ropivacaine 80 mg will be used
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: intrathecal infusion — morphine 150 mcg will be used by intrathecal administration
  Other Names: morphine
  Arms: morphine
Drug: Intravenous Infusion — tramadol administration
  Other Names: tramadol
  Arms: tramadol
Drug: Ropivacaine injection — bilateral transversus abdominis plane block by using ropivacaine 80 mg
  Other Names: transversus abdominis plane lock
  Arms: ropivacaine

SUMMARY:
investigators aim to compare the efficacy of intrathecal morphine, intravenous tramadol and transversus abdominis plane block in the treatment of catheter related bladder discomfort syndrome in patients scheduled for robotic assisted laparoscopic prostatectomy

DETAILED DESCRIPTION:
patients scheduled for robot assisted laparoscopic prostatectomy will be treated depending on the belonging group. In the morphine group patients will receive intrathecal morphine 0,15 mg; in the transversus abdominis plane block patients will receive ropivacaine 80 mg; in the tramadol group patients will receive intravenous continuous infusion of tramadol 400 mg for the first 24 hours postoperatively. All data will be collected in the post anesthesia room and in the ward until the first post operative day.

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for robotic assisted laparoscopic prostatectomy

Exclusion Criteria:

* coagulation disorders and platelet dysfunction for spinal arm
* obesity for transversus abdominis plane block arm
* left ventricular ejection fraction < 30%, end-stage renal disease and neurological disorders for all groups

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
catheter related bladder discomfort syndrome | immediately after surgery
  grade 0 to III

SECONDARY OUTCOMES:
pain relief | immediately after surgery
  assessment of post-operative pain by a 0 to 10 numeric rating score

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided